CLINICAL TRIAL: NCT01174862
Title: Comparative Cohort Study on the Outcome of Patients With Normal and Reduced Acetylsalicylic Acid Responsiveness Undergoing Coronary Artery Bypass Surgery
Brief Title: Aspirin Responsiveness and Outcome in Coronary Artery Bypass Graft (CABG) Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Daniel Bolliger, PD Dr. med. Daniel Bolliger, University Hospital, Basel, Switzerland
Other Study IDs: 288/09
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Bypass Graft Triple Vessel; Myocardial Ischemia; Thrombosis; Antithrombotic Drugs [Platelet-aggregation Inhibitors] Causing Adverse Effects in Therapeutic Use
Keywords: aspirin; aspirin responsiveness; long-term outcome; CABG
MeSH Terms: conditions — Myocardial Ischemia; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aspirin responder: Normal aspirin responsiveness in ASPI test (Multiplate)
- Aspirin non-responder: Reduced aspirin responsiveness in ASPI test (Multiplate)

SUMMARY:
In patients undergoing coronary artery bypass graft (CAGB) surgery, aspirin is commonly prescribed to prevent graft thrombosis and myocardial ischemia. However, there are still a significant number of grafts occluding in the postoperative period. This is partly attributed to reduced aspirin responsiveness, also called "aspirin resistance". At the moment, no standardized definition or laboratory test is available to quantify "aspirin resistance", and strong platelet reactivity in laboratory tests is not necessarily associated with increased thrombotic events. However, there is increasing evidence that reduced aspirin responsiveness in platelet function analyzers is associated with adverse long-term outcome and higher incidence of major adverse events in patients with stable coronary artery disease and in patients undergoing percutaneous coronary intervention. In patients undergoing coronary artery bypass graft surgery, the predictive value of a laboratory finding of reduced aspirin responsiveness remains unclear.

Therefore, the aim of this study is to prospectively evaluate whether the pre- and/or postoperative laboratory finding of reduced aspirin responsiveness defined by MultiplateTM platelet function analyzer is associated with higher incidences of adverse outcome after 30 days and 12 months in patients undergoing CABG surgery.

ELIGIBILITY:
Inclusion criteria:

* patient undergoing elective CABG surgery
* therapy with aspirin until at least 2 days before surgery
* written informed consent

Exclusion criteria:

* missing written consent
* no therapy with aspirin or therapy stopped more than 2 days before surgery
* therapy with clopidogrel more than 3 days before surgery
* emergency surgery
* surgery including more than CABG
* inborn or acquired platelet disorders
* therapy with Selective Serotonin reuptake inhibitors (SSRI)
* severe hepatopathy (spontaneous Quick <70%)
* severe kidney disease (creatinine clearance < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective CABG surgery (on-pump and off pump surgery)
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Death and/or major cardiac or thromboembolic events | 12 months after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bolliger, MD, Principal Investigator — Department of Anaesthesia and Intensive Care Unit, University Hospital Basel, Switzerland
Locations (1):
- Department of Anaesthesia and Intensive Care Unit, Univeristy Hospital Basel, Switzerland, Basel, Canton of Basel-City, Switzerland